CLINICAL TRIAL: NCT02718924
Title: Thromboelastometry (ROTEM) For Detecting Hypercoagulability in Morbidly Obese and Non Obese Parturients Following Cesarean Section Delivery: An Observational Study
Brief Title: Detecting Hypercoagulability in Morbidly Obese and Non Obese Parturients Following Cesarean Section Delivery
Status: Completed | Type: Observational
Sponsor: Corniche Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ch23031401
Record Dates: First submitted 2016-01-17; First posted 2016-03-24 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Pregnancy; Obesity; Hypercoagulability
Keywords: Thromboelastometry; pregnancy; obesity
MeSH Terms: conditions — Obesity; Thrombophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- morbidly obese pregnant: Term pregnant women with BMI more than 40
- non obese pregnant: Term pregnant women with BMI less than 30

SUMMARY:
Investigators hypothesized that the impact of surgery in terms of inducing a hypercoagulable state is more evident in morbidly obese pregnant women as opposed to their non-obese counterparts. The aim of this study is to investigate the change in coagulation status of morbidly obese and non-obese pregnant women following cesarean section delivery using thromboelastometry. This observational study would also make it possible to calculate the sample size for a future prospective controlled clinical trial to compare the incidence of Hypercoagulability in morbidly obese parturients as opposed to their non-obese counterparts. To the best of our knowledge, no other work has been done any in this area.

DETAILED DESCRIPTION:
Following institutional ethical committee approval, 20 morbidly obese (BMI>40) and 20 non-obese (BMI < 30) parturients undergoing elective low segment cesarean section (LSCS) delivery under spinal subarachnoid block will be recruited into the study. A written informed consent will be obtained from all parturients prior to inclusion. All patients will receive an information sheet at the preoperative assessment visit to inform them about this study. Patients with a history of past or current thromboembolism will be excluded from the study as well as those with liver disease and those already on anticoagulant/anti-platelet therapy for repeated miscarriage or other indications. History of thromboembolism is defined as an arterial or deep venous thrombosis, catheter thrombosis, or pulmonary embolism diagnosed by ultrasound or spiral computed tomography (CT). Preoperative baseline full blood count and clotting profile will be done. Parturients with abnormal platelet count or coagulation results and those who will need conversion to general anesthesia will be excluded.

Data and sample collection Preoperative BMI, co-existing morbidities and laboratory test results including INR, PTT and platelet count as well as operative time and postoperative clinical or radiological evidence of thromboembolism will be recorded. A blood sample will be collected for ROTEM analysis prior to establishing the block (baseline), immediately after surgery and 8 hours later.

ROTEM analysis

Coagulability will be assessed using the ROTEM thromboelastometry analyzer (The ROTEM® delta, Tem Systems Inc.®, Munich, Germany). Extrinsic rotational thromboelastometry (EXTEM), intrinsic rotational thromboelastometry (INTEM) and FIBTEM will be measured for each blood sample. Clotting time (CT), clot formation time (CFT) and maximum clot firmness (MCF) will be recorded. Total clot strength will be assessed by "G" value as calculated according to the formula: (5000xMCF)/100-MCF and expressed as dynes/cm2 . G has been shown to be valuable in diagnosing hypo- and hypercoagulability . In non-obstetric cohorts, hypercoagulability was defined as a G value of ≥ 11.7 dynes/cm2 and hypocoagulability as a G value of <5.0 dynes/cm2 (values provided by manufacturer).

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at term presenting for cesarean section under spinal anaesthesia with BMI less than 30 and more than 40

Exclusion Criteria:

* Patients with BMI between 30 and 40 BMI
* Patients with a history of past or current thromboembolism.
* Patients with history of liver disease and those on anticoagulant/anti-platelet therapy
* Patients who requires perioperative blood transfusion
* Patients having General anaesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Term pregnant women presenting for elective cesarean section under spinal anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Calculated clot strength using EXTEM Maximum Clot Firmness (G value for EXTEM) | 8 hours
  "G" value will be calculated according to the formula: (5000xMCF)/100-MCF and expressed as dynes/cm2

SECONDARY OUTCOMES:
EXTEM clotting time and clot formation time in seconds. | 8 hours
  measured ROTEM thromboelastometry variables
EXTEM maximum clot firmness in millimeters | 8 hours
  measured ROTEM thromboelastometry variable
INTEM clotting time and clot formation time in seconds. | 8 hours
  measured ROTEM thromboelastometry variables
INTEM maximum clot firmness in millimeters | 8 hours
  measured ROTEM thromboelastometry variable
FIBTEM maximum clot firmness in millimeters | 8 hours
  measured ROTEM variable

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Samy Abdel Raheem, FRCA, Principal Investigator — Consultant Anaesthetist; Tarek Ansari, FFARCSI, Principal Investigator — Consultant Anaesthetist; Waleed Riad, MD, Principal Investigator — Consultant Anaesthetist
Locations (1):
- Corniche Hospital, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
No plan